CLINICAL TRIAL: NCT02921022
Title: Pilot Study Of Gemcitabine, Nab-paclitaxel, PEGPH20 and Rivaroxaban for Advanced Pancreatic Adenocarcinoma
Brief Title: Study Of Gemcitabine, Nab-paclitaxel, PEGPH20 and Rivaroxaban for Advanced Pancreatic Adenocarcinoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Halozyme Therapeutics (Industry); Miami Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-1066
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Cancer; Advanced Pancreatic Ductal Adenocarcinoma
Keywords: Gemcitabine; Nab-paclitaxel; PEGPH20; Rivaroxaban; thromboembolic event (TE); 16-1066
MeSH Terms: conditions — Pancreatic Neoplasms; Thromboembolism | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; PEGPH20

ARMS (2):
- Patients without a prior thromboembolic event (TE) (Experimental): Patients without a prior TE will be treated with prophylactic dose and schedule of rivaroxaban (10 mg QD), together with standard dose and schedule of gemcitabine, nab-paclitaxel and PEGPH20.
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel; Drug: PEGPH20
- Patients with a prior thromboembolic event (TE) (Experimental): Patients with a prior TE will be treated with therapeutic dose and schedule of rivaroxaban (15 mg BID for 21 days for induction if indicated, then 20 mg QD for chronic treatment), together with standard dose and schedule of gemcitabine, nab-paclitaxel and PEGPH20.
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel; Drug: PEGPH20

INTERVENTIONS:
Drug: Gemcitabine
Drug: Nab-paclitaxel
Drug: PEGPH20

SUMMARY:
The purpose of this study is to test any good and bad effects of the study drug called PEGPH20. PEGPH20 alone is considered investigational. The Food and Drug Administration (FDA) has not approved the marketing or sale of PEGPH20, but have authorized its use in research studies with humans. PEGPH20 could shrink the cancer but it also can cause side effects. PEGPH20 is an enzyme that breaks down a specific tissue component called hyaluronan produced by some tumors. Pancreatic tumors often have a large amount of hyaluronan. The removal of hyaluronan from tumors may decrease tumor growth.

ELIGIBILITY:
Inclusion Criteria:

* Signed, written Institutional Review Board (IRB)-approved Informed Consent Form (ICF).
* Histologically confirmed locally advanced unresectable (Stage III) or Stage IV PDAC.
* Measurable or evaluable disease on computed tomography (CT) or magnetic resonance imaging (MRI) scan per RECIST v1.1.
* For patients with locally advanced disease, no previous radiotherapy, surgery, chemotherapy, or investigational therapy for the treatment of PDAC is permitted. For patients with metastatic disease, prior treatment for non-metastatic disease with 5-FU or gemictabine administered as radiation sensitizer, or as a cytotoxic therapy, in the adjuvant setting is allowed, provided at least 6 months have elapsed since completion of the last dose and no ≥ Grade 2 treatment-related toxicities are present.
* Karnofsky Performance Status ≥70%.
* Life expectancy ≥3 months.
* Age ≥18 years.
* A negative serum pregnancy test, if female of reproductive potential.
* Screening clinical laboratory values as follows, performed within 14 days prior to day 1:

  * Total bilirubin ≤1.5 times upper limit of normal (ULN).
  * Aspartate aminotransferase ([AST]; serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase ([ALT]; serum glutamic pyruvate transaminase [SGPT]) ≤2.5 times ULN, (if liver metastases are present, then ≤5 times ULN is allowed).
  * Serum creatinine ≤2.0 mg/dL or calculated creatinine clearance ≥60 mL/min.
  * Serum albumin ≥3.0 g/dL.
  * Absolute neutrophil count (ANC) ≥1,500 cells/mm3.
  * Platelet count ≥100,000 plt/mm3.
  * Hemoglobin ≥9 g/dL
  * Prothrombin time (PT)/international normalized ratio (INR) within normal limits (±15%) or within therapeutic range if on warfarin.
  * Partial thromboplastin time (PTT) within normal limits (±15%).
* For men and women of reproductive potential, agreement to use an effective contraceptive method from the time of screening and throughout their time on study. Effective contraceptive methods consist of prior sterilization, intra-uterine device, oral or injectable contraceptives, and/or barrier methods. Abstinence alone is not considered an adequate contraceptive measure for the purposes of this study.

Exclusion Criteria:

* Known central nervous system involvement or brain metastases.
* New York Heart Association Class III or IV cardiac disease or myocardial infarction within the past 12 months.
* Known, clinically significant carotid artery disease.
* Known, increased risk of bleeding.
* Patients with TE event occurring > 6months prior to enrollment and receiving active anticoagulation.
* Patients with any prior history of arterial thrombosis or symptomatic pulmonary embolism.
* Patients with current use of megestrol acetate (use with 10 days of Day 1) will be excluded.
* Active, uncontrolled bacterial, viral, or fungal infection requiring systemic therapy.
* Known active infection with human immunodeficiency virus, hepatitis B, or hepatitis C.
* Known allergy to hyaluronidase.
* Patients with prosthetic heart valves
* Women currently pregnant or breastfeeding.
* Intolerance of dexamethasone.
* History of another primary cancer within the last 3 years with the exception of non-melanoma skin cancer or curatively-treated cervical carcinoma in-situ.
* History of transient ischemic attack (TIA) or cerebrovascular accident (CVA).
* Any other disease, metabolic dysfunction, physical examination finding or clinical laboratory finding that leads to reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, that may affect the interpretation of the results, or that may render the subject at high risk for treatment complications.
* Other unspecified reasons that, in the opinion of the Investigator, make the subject unsuitable for the study.
* Inability to comply with study and follow-up procedures as judged by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-10; Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
rate of symptomatic TE events | 1 year
  This includes any grade 2 or grade 3 thromboembolic event as defined by NCI CTCAE v4.0 found on incidental imaging, which would indicate a need for medical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Yu, MD, MSc, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Hartford Healthcare Cancer Institute @ Hartford Hospital, Hartford, Connecticut
  - Miami Cancer Institute, Miami, Florida
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/